CLINICAL TRIAL: NCT02641509
Title: Accuracy in Resection of Non-pedunculated Colonic Lesions 5-20 mm With/Without Using NBI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Alida Andrealli, MD, Valduce Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 854/2015
Record Dates: First submitted 2015-11-30; First posted 2015-12-29 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Polypectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NBI to perform the polipectomy (Experimental): this arm will undergo polypectomy with the use of NBI to define the margins of the lesion
  Interventions: Device: NBI during polypectomy
- no NBI to perform the polypectomy (Experimental): this arm will undergo polipectomy without the use of NBI to define the margins of the lesion
  Interventions: Device: no NBI during polypectomy

INTERVENTIONS:
Device: NBI during polypectomy — NBI to perform the polipectomy
  Arms: NBI to perform the polipectomy
Device: no NBI during polypectomy — no NBI to perform the polypectomy
  Arms: no NBI to perform the polypectomy

SUMMARY:
Interval colon cancers are an important clinical issue. A recent paper from Pohl et al focused on non-pedunculated polyps of 5-20 mm, evaluating non complete polypectomy revealing that 10% of these polyps were not completely resected. This fact was attributed to size and histology. In this study the investigators want to evaluate the radical resection of non-pedunculated polyps of 5-20 mm by performing biopsies on the margins immediately after polypectomy, to establish if the use of Narrow Band Imaging (NBI) could be useful in the definition of the margins of the lesion before polypectomy.

DETAILED DESCRIPTION:
Interval colon cancers are an important clinical issue. Literature dealing with technics and quality of polypectomy is scarce. A recent paper from Pohl et al focused on non-pedunculated polyps of 5-20 mm, evaluating non complete polypectomy and factors related to it, revealing that 10% of these polyps were not completely resected. This fact was attributed to size and histology (the majority of non completely resected ones, were polyps of 10-20 mm and with serrated characteristics at the histology). In this study the investigators want to evaluate the radical resection of non-pedunculated polyps of 5-20 mm by performing biopsies on the margins immediately after polypectomy, to establish if the use of Narrow Band Imaging (NBI) could be useful in the definition of the margins of the lesion before polypectomy.

ELIGIBILITY:
Inclusion Criteria:

* Every polyp ≥ 5 mm and ≤ 20 mm

Exclusion Criteria:

* Inflammatory bowel Disease and/or International Normalized Ratio > 1.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2016-01; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
NBI efficacy in predicting radicality of polypectomy by taking random biopsies of margins after resection of the lesion | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Valduce Hospital, Como, Italy